CLINICAL TRIAL: NCT06171867
Title: Preterm Neonate/ Neonatal Embedded Universal Microelectronic Wearable Acquisition for Cardio Respiratory Intensive Therapy. Clinical Assessment of Device Usability and Reliability
Brief Title: PNEUMACRIT Device for Neonatal Cardio Respiratory Monitoring
Acronym: PNEUMACRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Middlesex University (Other)
Responsible Party: Principal Investigator, Merja Kallio, MD, PhD, Principal investigator, Associate professor of pediatrics, University of Oulu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EETTMK: 73/2021
Record Dates: First submitted 2023-11-23; First posted 2023-12-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Neonatal Respiratory Distress
Keywords: Electrical impedance tomography, neonate
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: The device feasibility will be assessed in clinical environment with feedback from both the patient parents and nurses in NICU/PICU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility of the PNEUMACRIT belt (Experimental): Neonates will be monitored with a PNEUMACRIT electrode belt for 6 to 24 hours. After the study period, patient parents and nurses will give feedback.
  Interventions: Device: PNEUMACRIT

INTERVENTIONS:
Device: PNEUMACRIT — Monitoring of breathing

SUMMARY:
The usability of a new PNEUMACRIT system is studied in clinical environment in this feasibility study.

DETAILED DESCRIPTION:
Electrical impedance tomography is a noninvasive monitoring tool for neonatal lung aeration and breathing. This feasibility study will assess the usability of a new PNEUMACRIT electrode belt in clinical environment.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient at Oulu University Hospital PICU or NICU
* Gestational age at birth over 32 weeks
* Weight 2000-5000g
* Postnatal age > 12 hours
* Written informed consent from the parents of legal representative
* Non-invasive monitoring of oxygen saturation and ECG

Exclusion Criteria:

* Postmenstrual age < 32 weeks
* Weight at time of the study < 2000g or > 5000g
* Chest skin lesion preventing safe use of the electrode belt
* Recent chest surgery within the past 7 days (e.g. thoracotomy)

Ages: 12 Hours to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Proportion (%) of recording time with high quality EIT-signal | 6-24 hours
  Proportion of time that the collected EIT signal is accurate enough for reliable image reconstruction and observations of changes in lung aeration

SECONDARY OUTCOMES:
Staff and parent questionnaires | 48 hours
  After the study period, the patient parents and nurses will give feedback on the device and its feasibility with a structured questionnaire including also free text fields

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.pneumacrit.com/